CLINICAL TRIAL: NCT07187167
Title: Efficacy and Safety of the RD Regimen (Lenalidomide, Dexamethasone) in the Treatment of Rosai-Dorfman Disease: A Prospective, Multicenter, Single-Arm Study.
Brief Title: Efficacy and Safety of the RD Regimen(Lenalidomide, Dexamethasone) for Rosai-Dorfman Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH005
Record Dates: First submitted 2025-08-25; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Rosai-Dorfman Disease
MeSH Terms: conditions — Histiocytosis, Sinus | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, interventional study, with a planned number of subjects: approximately 40 cases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with RDD (Experimental): Patients with RDD who are treatment-naive or have not previously received lenalidomide; aged 18-80 years; ECOG PS 0-2.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — The combination therapy period consists of 12 cycles: Lenalidomide: 25mg, orally, D1-21, every 28 days per cycle. Combined with Dexamethasone: 40mg, orally, D1, 8, 15, 22, every 28 days per cycle. The single-agent maintenance period consists of 12 cycles: Lenalidomide: 25mg, orally, D1-21, every 28 days per cycle. The total treatment duration is 24 cycles or until disease progression, death, or the occurrence of intolerable toxicity.
  Other Names: INNs
Drug: Dexamethasone — The combination therapy period consists of 12 cycles: Lenalidomide: 25mg, orally, D1-21, every 28 days per cycle. Combined with Dexamethasone: 40mg, orally, D1, 8, 15, 22, every 28 days per cycle. The single-agent maintenance period consists of 12 cycles: Lenalidomide: 25mg, orally, D1-21, every 28 days per cycle. The total treatment duration is 24 cycles or until disease progression, death, or the occurrence of intolerable toxicity.
  Other Names: INNs

SUMMARY:
In patients with Rosai-Dorfman disease (RDD), a treatment regimen of lenalidomide combined with dexamethasone is planned to be used.

DETAILED DESCRIPTION:
Patients received oral lenalidomide 25mg on days 1-21 and dexamethasone 40mg on days 1, 8, 15, 22, in 28-day cycles for 12 total cycles.

ELIGIBILITY:
Inclusion Criteria:

* Definitively diagnosed adult RDD patients;
* Aged between 18 and 80 years;
* Treatment-naive or refractory/relapsed;
* ECOG performance status score ≤ 2;
* Judged by clinicians as suitable for treatment with this protocol;
* Patients or their families able to understand the study protocol and willing to participate in the study, providing written informed consent.

Exclusion Criteria:

* Subjects who have undergone major surgery within 4 weeks prior to the first dose of the study;
* Subjects who have received radiotherapy within 4 weeks prior to the first dose of the study;
* Subjects with a history of myocardial infarction within the past year;
* Patients with New York Heart Association (NYHA) Class 3 or 4 congestive heart failure, or a history of NYHA Class 3 or 4 congestive heart failure;
* Pregnant or lactating women;
* Patients who cannot strictly practice contraception after participating in the study;
* Abnormal liver and kidney function: creatinine level ≥176.8 μmol/L (2 mg/dL), transaminase and bilirubin levels more than 2 times the upper limit of normal
* Abnormal blood counts: absolute neutrophil count less than 1×10^9/L, platelet count less than 50×10^9/L;
* Patients or their families who cannot understand the conditions and objectives of the study;
* Any other situation where the investigator considers the patient unsuitable to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2027-04-12 (Estimated); Study Completion 2027-04-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time （PFS) | From enrollment to the end of treatment at 8 weeks
  PFS defined as the time from RD initiation to first documented disease progression, relapse after RD, death from any cause, or last follow-up.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From enrollment to the end of treatment at 8 weeks
  The overall response rate (ORR) was defined as the cumulative proportion of patients attaining either a complete response (CR) or partial response (PR) .
Overall Survival (OS) | From enrollment to the end of treatment at 8 weeks"
  OS was measured from RD start to death or last follow-up
Adverse events | From enrollment to the end of treatment at 8 weeks
  Toxicities were recorded and graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

OTHER OUTCOMES:
Correlation between next-generation sequence (NGS) and therapeutic efficacy/PFS | From enrollment to the end of treatment at 8 weeks"
  Correlation between the positivity of NGS in MAPK pathway and therapeutic efficacy/PFS
Fact-G | From enrollment to the end of treatment at 8 weeks
  The score of Functional Assessment of Cancer Therapy - General

CONTACTS AND LOCATIONS:
Overall Officials: Xinxin XX Cao, doctor, Study Chair — NCC, CICAMS
Locations (1):
- Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No